CLINICAL TRIAL: NCT06395545
Title: Evaluation of the Efficacy of an Electronic Constant-speed Injector in Reducing Infusion Pain Associated With Local Infiltrative Anesthesia in a Scalp Surgery
Brief Title: Local Anesthesia and Electronic Injector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Chong Hyun Won, Dermatology professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2022-1463
Record Dates: First submitted 2024-04-26; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Hair Diseases
MeSH Terms: conditions — Hair Diseases

STUDY DESIGN:
Intervention Model Description: This study was a single-blind, randomized, controlled trial. We enrolled patients who underwent local infiltrative anesthesia in an area >5 cm during scalp surgery at Dr. Hwang's Hair Clinic, Seoul, Korea, between March 2022 and August 2022.
Masking Description: The injection site in a patient was divided into two sides (left and right). The method of local infiltration (manual or using the electronic injector) was randomly assigned to each side of the surgical field, and 2.5 cc (0.5 cc at five separate areas) of local anesthetic was injected individually using a 5 cc syringe with a 31-gauge needle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants ( control and test group ) (Experimental): At room temperature, 1% lidocaine combined with 1:100,000 epinephrine was used as a local anesthesia. The electronic constant-speed injector, i-JECT® (MediHub Inc., Gyeonggi-do, Korea) (Figure 1) was used, and the injection speed of the injector was set at level 1 (0.25 mL/s) or level 2 (0.4 mL/s). The injection site in a patient was divided into two sides (left and right). The method of local infiltration (manual or using the electronic injector) was randomly assigned to each side of the surgical field, and 2.5 cc (0.5 cc at five separate areas) of local anesthetic was injected individually using a 5 cc syringe with a 31-gauge needle. All injections were administered by a single surgeon (Sung Joo Tommy Hwang) to reduce inter-operator variation.
  Interventions: Device: Electronic injector

INTERVENTIONS:
Device: Electronic injector — At room temperature, 1% lidocaine combined with 1:100,000 epinephrine was used as a local anesthesia. The electronic constant-speed injector, i-JECT® (MediHub Inc., Gyeonggi-do, Korea) (Figure 1) was used, and the injection speed of the injector was set at level 1 (0.25 mL/s) or level 2 (0.4 mL/s). The injection site in a patient was divided into two sides (left and right). The method of local infiltration (manual or using the electronic injector) was randomly assigned to each side of the surgical field, and 2.5 cc (0.5 cc at five separate areas) of local anesthetic was injected individually using a 5 cc syringe with a 31-gauge needle. All injections were administered by a single surgeon (Sung Joo Tommy Hwang) to reduce inter-operator variation.

SUMMARY:
Local anesthesia-related pain is associated with injection speed. An electronic constant-speed injector was developed for slow and steady injection to alleviate dermatological anesthesia pain. The investigators aimed to validate the efficacy of an electronic constant-speed injector in reducing pain during local infiltrative anesthesia by comparing it to the conventional manual injection method. Patients who underwent local infiltrative anesthesia in an area >5 cm during scalp surgery were selected. Each side of the surgical field was randomly assigned a manual or electronic injector for local infiltration. Each participant used the numeric rating scale (NRS) to rate infiltration-related pain on each side.

DETAILED DESCRIPTION:
Local anesthesia (LA) is an imperative component of dermatologic surgery. It allows large procedures to be performed comfortably even in an office setting. However, if patients undergo painful anesthesia injection, this may negatively affect their overall experience regarding dermatologic procedures.

Therefore, numerous studies have been conducted on LA-related pain reduction. Buffering or warming local anesthesia, administering topical anesthesia or cooling anesthesia, and distracting patients with stimuli such as vibration or music are discussed to be helpful for relatively painless LA. Furthermore, low speed of injection is suggested as one of the methods to alleviate infusion-induced pain which refers to the pain associated with the infiltration of anesthetic fluid into the tissue. However, speed control with manual injection is challenging. Therefore, "computer-controlled local anesthetic delivery (CCLAD) devices" have been developed to inject LA into the tissues at a set speed. A computer-controlled local anesthetic delivery device aims to reduce LA-related pain through slow injection. The first CCLAD, Wand (Milestone Scientific Inc., Livingston, USA), was introduced in 1997 in dentistry. These CCLAD systems have been predominantly investigated in dentistry, but are also expected to relieve LA-related pain in various dermatological procedures. However, no objective study has been conducted about the efficacy of an electronic constant-speed injector in decreasing local anesthetic pain in dermatology.

Therefore, the investigators aimed to confirm the efficacy of an electronic constant-speed injector in pain reduction during local infiltrative anesthesia in a scalp surgery of dermatologic fields by comparing it to the conventional manual injection method.

This study was a single-blind, randomized, controlled trial. The investigators enrolled patients who underwent local infiltrative anesthesia in an area >5 cm during scalp surgery at Dr. Hwang's Hair Clinic, Seoul, Korea, between March 2022 and August 2022.

At room temperature, 1% lidocaine combined with 1:100,000 epinephrine was used as a local anesthesia. The electronic constant-speed injector, i-JECT® (MediHub Inc., Gyeonggi-do, Korea) (Figure 1) was used, and the injection speed of the injector was set at level 1 (0.25 mL/s) or level 2 (0.4 mL/s). The injection site in a patient was divided into two sides (left and right). The method of local infiltration (manual or using the electronic injector) was randomly assigned to each side of the surgical field, and 2.5 cc (0.5 cc at five separate areas) of local anesthetic was injected individually using a 5 cc syringe with a 31-gauge needle. All injections were administered by a single surgeon (Sung Joo Tommy Hwang) to reduce inter-operator variation.

Regarding the training of the participants, a short clip explaining the forthcoming procedures and related pain were introduced to the participants and the informed consents were obtained. NRS ranging from 0 (painless) to 10 (worst pain possible) was used as an objective tool for pain evaluation. Participants used a numeric rating scale (NRS) to rate their level of infusion-related pain immediately after receiving each 0.5 cc injection of local anesthesia.

Statistical analysis was performed using IBM SPSS (ver. 21.0; IBM Corp., Armonk, NY, USA). A paired-sample t-test was used to identify whether the NRS score of manual injection was higher than that of mechanical injection. Independent-sample t-test was used to assess for differences in the efficacy of injectors between sexes. P < 0.05 was considered to be statistically significant.

This study was approved by the institutional review boards of Asan Medical Center (2022-1463) and was conducted according to the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Participants who underwent local infiltrative anesthesia in an area >5 cm during scalp surgery at Dr. Hwang's Hair Clinic, Seoul, Korea, between March 2022 and August 2022

Exclusion Criteria:

* Participants who did not consent to the study enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | During the intervention
  a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea